CLINICAL TRIAL: NCT04603729
Title: Comparison of Efficacy of Dexamethasone and Methylprednisolone in Moderate to Severe Covid 19 Disease
Acronym: covid19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Syeda Arzinda Fatima, Assistant Professor, Fatima Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMH-06-2020-IRB-763-M
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Covid 19 Disease
Keywords: covid19; dexamethasone; methlprednisolone; corticosteroids
MeSH Terms: conditions — COVID-19 | interventions — Dexamethasone; Calcium Dobesilate; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 dexamethasone (Active Comparator): participants will receive dexamethasone 8mg/day Intravenous for 5 days
  Interventions: Drug: Dexamethasone 2 MG/ML
- group 2 methylprednisolone (Active Comparator): participants will receive methylprednisolone 1mg/kg/day intravenous for 5 days
  Interventions: Drug: Methylprednisolone Injection

INTERVENTIONS:
Drug: Dexamethasone 2 MG/ML — Dexamethasone 8mg/day will be given intravenous for 5 days to group 1 participants
  Other Names: decadron
  Arms: group 1 dexamethasone
Drug: Methylprednisolone Injection — methylprednisolone 1mg/kg/day will be given intravenous for 5 days to group 2 participants
  Other Names: solumedrol
  Arms: group 2 methylprednisolone

SUMMARY:
The investigator will select participants with moderate to severe covid 19 disease admitted in Fatima memorial hospital. The investigator will divide them in two groups according to convenience sampling. Group 1 will be given dexamethasone 8mg/day and group 2 will be given methylprednisolone 1mg/kg/day IV for 5 days. The investigator will compare the improvement in temperature, oxygen requirement and CRP level at day zero and day 5 in both the groups.

DETAILED DESCRIPTION:
The investigators enrolled first 100 participants admitted in covid unit of Fatima memorial hospital who fulfilled the inclusion criteria and signed informed consent. Baseline oxygen saturation and clinical findings were noted. Chest x-ray was done on admission. Baseline labs were sent, initial level of CRP (C-reactive protein) was noted down.

Patients with oxygen saturation < 94% on room air with normal chest x-ray and CRP between 30 - 50, were labelled as having moderate covid 19 disease. Patients with CRP> 50 and having infiltrates on chest x-ray at the time of admission were considered having severe covid 19 disease. Intravenous methylprednisolone in a dose of 1 mg/kg/day in 2 divided doses or dexamethasone 8 mg/day IV was given to alternate patients for 5 days. After 5 days, the investigator again recorded the oxygen saturation, CRP level and repeat chest x-ray findings.

Patients were given tocilizumab and convalescent plasma as and when indicated. Oxygen was given by nasal cannula and face mask. Patient was shifted to ICU if clinical condition deteriorated and/or mechanical ventilation is needed.

The investigator noted the improvement in clinical, radiological and biochemical parameters of the patient on day 0 that is admission day and later on day 5 after giving steroids (methylprednisolone or dexamethasone) for 5 days.

Data was analyzed using SPSS version 25.0. Descriptive statistics like frequency and means were calculated. Paired sample t-test was applied for comparison of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Covid PCR positive
3. Patient having oxygen saturation < 94% on room air, regardless of chest x-ray findings
4. Moderate or severe covid 19 disease according to operational definition.
5. Patients who sign informed consent.

Exclusion Criteria:

1. Severe immunosuppression like HIV( Human immunodeficiency Virus) or long term use of immunosuppressant for any other chronic illness
2. Patients who need corticosteroids for any other disease like asthma, rheumatoid arthritis.
3. Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
temperature (F) | 5 days
  reduction in temperature in degree farrenheit
oxygen saturation(%) | 5 days
  reduction in oxygen requirement in lit/min
CRP (mg/dl) | 5 days
  mean reduction in CRP mg/dl in 5 days
mortality | 5 days
  number of patients died
ICU transfer | 5 days
  number of patients shifted to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid A Khan, MBBS, FACM, Study Chair — Fatima Memorial Hospital; Arzinda F Syeda, MBBS, FCPS, Principal Investigator — Fatima Memorial Hospital
Locations (1):
- Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
patient name and medical record will be confidential, onle the principal investigator will have access to data. Results of study will be shared with other researchers